CLINICAL TRIAL: NCT05905276
Title: ERAS for Ambulatory TURBT: Enhancing Bladder Cancer Care (EMBRACE) Randomized Controlled Trial Protocol
Brief Title: Enhanced Recovery After Surgery (ERAS) for Ambulatory TURBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00392063
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Bladder Cancer
Keywords: ERAS; Ambulatory Surgery; Quality of Recovery; Quality of Care; Bladder Cancer; Patient-centered outcomes; Enhanced Recovery after Surgery
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Patients in the usual care arm of the trial will experience the present-day care pathway of ambulatory TURBT at Johns Hopkins Hospital.
  Interventions: Other: Standard of Care
- ERAS Protocol (Experimental): The ERAS protocol for ambulatory TURBT has been designed based on patient and provider input, a needs assessment of 150 patients in the hours after TURBT, a review of the literature, and experience with other ambulatory ERAS protocols already implemented at Johns Hopkins Hospital. The ERAS protocol for ambulatory TURBT aims to optimize care delivered in the pre, intra and postoperative settings.
  Interventions: Other: ERAS Protocol

INTERVENTIONS:
Other: ERAS Protocol — The ERAS protocol for ambulatory TURBT has been designed based on patient and provider input, a needs assessment of 150 patients in the hours after TURBT, a review of the literature, and experience with other ambulatory ERAS protocols already implemented at Johns Hopkins Hospital. The ERAS protocol for ambulatory TURBT aims to optimize care delivered in the pre, intra and postoperative settings.
  Arms: ERAS Protocol
Other: Standard of Care — Patients in the usual care arm of the EMBRACE trial will experience the present-day care pathway of ambulatory TURBT at Johns Hopkins Hospital.
  Arms: Standard of Care

SUMMARY:
This is a single-center, randomized-controlled trial to investigate the effectiveness of an ERAS protocol compared to usual care in patients with bladder cancer undergoing ambulatory TURBT. The ERAS protocol is comprised of pre, intra and postoperative components designed to optimize each phase of perioperative care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected or known bladder cancer
* Age >= 18 years
* Undergoing initial or repeat TURBT
* Ambulatory TURBT with same day discharge home planned

Exclusion Criteria:

* Undergoing a planned concomitant procedure
* Inability to consent for themselves
* Unable to complete telephone-based follow up after discharge home
* Undergoing active treatment for muscle-invasive bladder cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-12-03 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Change in quality of recovery as assessed by Quality-of-Recovery 15 Scores (QoR-15) | Measured at enrollment through study completion, an average of 7 days.
  The QoR-15 score is a validated 15-item questionnaire that assesses quality of recovery in five dimensions: pain, physical comfort, functional autonomy, emotions, and psychological support. Each item is scored 0 to 10 with higher scores representing superior quality of recovery. The QoR-15 score is patient-reported outcome measure and has been extensively used to evaluate ERAS for both inpatient and ambulatory surgeries. It is a shorter and more patient-friendly version of the QoR-40 with equivalent psychometric properties.

SECONDARY OUTCOMES:
Change in lower urinary tract symptoms as assessed by the Urinary Tract Infection-Symptom and Impairment Questionnaire (UTI-SIQ-8) | Measured at enrollment through study completion, an average of 7 days.
  The UTI-SIQ-8 is a validated questionnaire of voiding symptom severity and bother, with higher scores representing worse symptoms (8-40).
Change in quality of life for bladder cancer patients as assessed by the Bladder Utility Symptom Scale (BUSS) | Measured at enrollment through study completion, an average of 7 days.
  Bladder Utility Symptom Scale - a validated 10-question instrument designed specifically for patients with bladder cancer, will be used to measure health-related quality of life (0-100), with higher scores representing higher quality of life.
Change in Pain as assessed by Visual Analogue Scale | Measured at enrollment through study completion, an average of 7 days.
  Dysuria, Suprapubic/Bladder, Urethral, Penis or Vulvar Pain Rated from 0 (No pain) to 10 (Unbearable pain)
Change in patient satisfaction as assessed by patient self-report | Measured at enrollment through study completion, an average of 7 days.
  Self-reported on a scale of 1 (lowest satisfaction) to 10 (highest satisfaction).
Change in degree of hematuria as assessed by patient self-report | Measured at enrollment through study completion, an average of 7 days.
  None, Pink, Red, Red with Clots as self-reported by patients
Change in incontinence | Average daily pad use measured at enrollment Measured at enrollment through study completion, an average of 7 days.
  Change in incontinence will be assessed by the average number of pads used per day
Change in opioid consumption | Measured at enrollment through study completion, an average of 7 days.
  Change in opioid consumption (Morphine milligram equivalents) obtained from medical record
Healthcare utilization | Measured at enrollment through study completion, an average of 30 days.
  Number of unplanned post-procedural ambulatory visits, emergency department visits, phone calls, and electronic messages assessed individually.
Complications as assessed by Clavien-Dindo complications | Measured at enrollment through study completion, an average of 30 days.
  Surgical complications as classified by Clavien-Dindo category.

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Rezaee, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rezaee ME, Mahon KM, Trock BJ, Nguyen TE, Smith AK, Hahn NM, Patel SH, Kates M. ERAS for Ambulatory TURBT: Enhancing Bladder Cancer Care (EMBRACE) randomised controlled trial protocol. BMJ Open. 2024 Jun 10;14(6):e076763. doi: 10.1136/bmjopen-2023-076763. PMID 38858157